CLINICAL TRIAL: NCT06254534
Title: Effect of Lidocaine, Dexmedetomidine, Esmolol and Magnesium Use on Optic Nerve Sheath Diameter and Hemodynamic Response After Laryngoscopy: Randomized, Controlled, Double-blind Trial
Brief Title: Lidocaine, Dexmedetomidine, Esmolol and Magnesium Effect on Optic Nerve Sheath Diameter After Laryngoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 106-2021
Record Dates: First submitted 2024-01-22; First posted 2024-02-12 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-06

CONDITIONS: Intracranial Hypertension; Endotracheal Intubation; Optic Nerve Sheath Diameter; General Anesthesia
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Intervention Model Description: Standardized, controlled, randomized, double blind
Who Masked: Participant, Investigator
Masking Description: The anesthesiology technician selected an envelope in order of numbers written on it and prepared unlabeled saline infusions according to the predetermined protocols of each group. Each group received one of the protocols as lidocaine (1.5 mg/kg), dexmedetomidine (1 mcg/kg), esmolol (1 mcq/kg), and magnesium (20 mg/kg) prepared in 50 ml of unlabeled physiological saline, after standard monitoring on the operating room table. In the control group, only saline was administered intravenously for 10 minutes; then general anesthesia was applied. Along with the study participants, the primary investigator was kept blind to the study groups as the sole applier of the ONSD measurement and the only observer of the hemodynamic changes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (Placebo Comparator): In the control group, only unlabeled saline prepared in 50 ml will be administered intravenously for 10 minutes before general anesthesia induction after standard monitoring on the operating room table.
  Interventions: Diagnostic Test: optic nerve ultrasonography
- Lidocaine (Experimental): lidocaine (1.5 mg/kg) within unlabeled saline prepared in 50 ml will be administered intravenously for 10 minutes before general anesthesia induction after standard monitoring on the operating room table.
  Interventions: Diagnostic Test: optic nerve ultrasonography
- magnesium (Experimental): magnesium (20 mg/kg) within unlabeled saline prepared in 50 ml will be administered intravenously for 10 minutes before general anesthesia induction after standard monitoring on the operating room table.
  Interventions: Diagnostic Test: optic nerve ultrasonography
- dexmedetomidine (Experimental): Dexmedetomidine (1 mcg/kg) within unlabeled saline prepared in 50 ml will be administered intravenously for 10 minutes before general anesthesia induction after standard monitoring on the operating room table.
  Interventions: Diagnostic Test: optic nerve ultrasonography
- Esmolol (Experimental): Esmolol (1 mcq/kg) within unlabeled saline prepared in 50 ml will be administered intravenously for 10 minutes before general anesthesia induction after standard monitoring on the operating room table.
  Interventions: Diagnostic Test: optic nerve ultrasonography

INTERVENTIONS:
Diagnostic Test: optic nerve ultrasonography — The primary investigator measured ONSD at times: first after anesthesia induction before laryngoscopy, second just after laryngoscopy, third five minutes after, and fourth ten minutes after intubation by ultrasound guidance with a high-frequency linear probe at T2 ophthalmic preset.

SUMMARY:
This clinical trial aims to compare the effects of lidocaine, dexmedetomidine, esmolol, and magnesium on optic nerve sheath diameter and hemodynamic response to laryngoscopy.

The participants will be patients determined to need intubation and general anesthesia for any elective surgery. Each participant will receive either lidocaine, dexmedetomidine, esmolol, magnesium, or none before anesthesia induction, according to randomization. The investigator will measure the optic nerve sheath diameter by ultrasonography before and after intubation. Researchers will compare the difference between optic nerve sheath diameter, systolic blood pressure, and heart rate before and after laryngoscopy and search for the most stable group. The trial aims to determine a general anesthesia induction protocol for patients sensitive to intracranial pressure changes reflected as optic nerve sheath diameter for easy monitoring.

DETAILED DESCRIPTION:
Laryngoscopy and endotracheal intubation could have detrimental effects on patients with limited physiologic reserve to cope with the possible hemodynamic alterations caused by the sympathoadrenal response. Although it is known to be a short-lasting and reversible physiological alteration, it could lead to more profound destructive effects, especially in patients with possible elevated intracranial pressure, such as in multi-trauma or intracranial hemorrhage. Therefore, minimizing alterations due to general anesthesia induction and intubation has been essential to optimize qualified critical patient management. Various drugs through different routes have been studied, focusing on hemodynamic alterations. However, as the health services and capabilities of the anesthesiologists improve, changes in outcome measures, such as intracranial pressure, could be observed directly by the integration of optic nerve ultrasonography (ONUS) as a part of point of care ultrasonographic (POCUS) examination. Notably, the measurement of optic nerve sheath diameter (ONSD) has been proven to be related to intracranial pressure, and several studies have even presented cut-off values with high diagnostic accuracy for increased intracranial pressure. Therefore, investigating ONSD during endotracheal intubation is a non-invasive, time and cost-effective method to observe the precise effects of drugs that can establish stability during intubation.

In this study, a wide variety of drugs from previous literature, lidocaine, dexmedetomidine, esmolol, and magnesium, has been chosen for their possible effectiveness in abolishing hemodynamic response to laryngoscopy. The study aims to compare the direct effect of these alternatives on ONSD during endotracheal intubation with concomitant hemodynamic changes. This study would like to emphasize POCUS and support the incorporation of ONUS as a valuable practice to improve general anesthesia management for fragile patients.

METHODS The trial design is a double-blind, randomized controlled study with the approval of our Institutional ethics committee (dossier no: 106-2021). The participants were assessed within patients scheduled for any elective surgery needing endotracheal intubation after January 2024 for eligibility. After obtaining written informed consent, 100 patients (Five groups; 1:1 distribution; n=20) were allocated, and the study was conducted in a tertiary care hospital with the principles outlined in the Helsinki Declaration.

Patients eligible for inclusion in this study are those aged 18 to 80 years who have undergone endotracheal intubation for general anesthesia and have an American Society of Anesthesiologists (ASA) Physical Status classification of I to III.

Patients are excluded if they had one of the following criteria: Patients allergic to dexmedetomidine, esmolol, lidocaine, magnesium; patients with uncontrolled hypertension or advanced heart failure with EF below 35%; patients with cardiac arrhythmia, especially Type 2 and 3 blocks, supraventricular arrhythmias, patients with renal failure (GFR below 30) or severe liver failure; patients with known acute or previous intracranial pathology and known diagnosis of epilepsy, predefined complex airway examination, patients who required more than one attempt at intubation or total laryngoscopy took more than 20 s.

Patient randomization and blindness Randomization will be performed using a computer-based algorithm in a 1:1 ratio into five (n= 20) named Groups A, B, C, D, and E and sealed into opaque envelopes by the study's primary investigator. The anesthesiology technician will select an envelope in order of numbers written on it and prepare unlabeled saline infusions according to the predetermined protocols of each group. Each group will receive one of the protocols as lidocaine (1.5 mg/kg), dexmedetomidine (1 mcg/kg), esmolol (1 mcq/kg), and magnesium (20 mg/kg) prepared in 50 ml of unlabeled physiological saline, after standard monitoring on the operating room table. In the control group, only saline will be administered intravenously for 10 minutes; then, general anesthesia will be applied. Along with the study participants, the primary investigator (B.C.) will be blind to the study groups as the sole applier of the ONSD measurement and the only observer of the hemodynamic changes.

All patients will receive standardized general anesthesia with 2 mg/kg propofol (Lipuro, Braun), 2 mcg/kg fentanyl (Talinat, VEM), 0,8 mg /kg rocuronium (Esmeron, Alessandroorsini) followed by 1 MAC sevoflurane (Sevorane, Abbott) in an air-oxygen mixture for maintenance of anesthesia with bi-spectral index monitorization (BIS, Medtronic). All endotracheal intubations will be done by practitioners with over two years of experience as anesthesiologists 2 min after the end of the rocuronium injection. The starting mechanical ventilator settings were volume-controlled ventilation with a positive end-expiratory pressure value of 5 mmHg for at least ten minutes.

The primary investigator (B.C.) will measure ONSD at times: first after anesthesia induction before laryngoscopy, second just after laryngoscopy, third five minutes after, and fourth ten minutes after intubation by ultrasound guidance with a high-frequency linear probe at T2 ophthalmic preset. Concurrently, systolic and mean blood pressure, heart rate, BIS, and end-tidal carbon dioxide will be recorded with the addition of peak pressures after intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years who will receive endotracheal intubation for general anesthesia and have an American Society of Anesthesiologists (ASA) Physical Status classification of I to III.

Exclusion Criteria:

* Patients allergic to dexmedetomidine, esmolol, lidocaine, and magnesium; patients with uncontrolled hypertension or advanced heart failure with EF below 35%; patients with cardiac arrhythmia, especially Type 2 and 3 blocks, supraventricular arrhythmias. Patients with renal failure (GFR below 30) or severe liver failure; patients with known acute or previous intracranial pathology and known diagnosis of epilepsy, predefined difficult airway examination. Patients who required more than one attempt at intubation or total laryngoscopy took more than 20 seconds.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
optic nerve sheath diameter | throughout the anesthesia
  optic nerve sheath ultrasonography will be used to measure optic nerve sheath diameter with a high-frequency linear probe at T2 ophthalmic preset at a distance of 3 mm from the posterior globe

SECONDARY OUTCOMES:
mean arterial pressure | throughout the anesthesia
  mean arterial pressure will be recorded at times of optic nerve sheath measurements
heart rate | throughout the anesthesia
  heart rate will be recorded at times of optic nerve sheath measurements

CONTACTS AND LOCATIONS:
Overall Officials: Berna Caliskan, Principal Investigator — Anesthesiology and Reanimation Department
Locations (1):
- Haseki Trainig and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berhanu D, Ferreira JC, Abegao Pinto L, Aguiar de Sousa D, Lucas Neto L, Tavares Ferreira J. The role of optic nerve sheath ultrasonography in increased intracranial pressure: A systematic review and meta analysis. J Neurol Sci. 2023 Nov 15;454:120853. doi: 10.1016/j.jns.2023.120853. Epub 2023 Oct 30. PMID 37925899
- [Background] Sriramka B, Warsi ZH, Sahoo J. Effects of adding dexmedetomidine to nebulized lidocaine on control of hemodynamic responses to laryngoscopy and intubation: A randomized clinical trial. J Anaesthesiol Clin Pharmacol. 2023 Jan-Mar;39(1):11-17. doi: 10.4103/joacp.JOACP_93_21. Epub 2022 Feb 10. PMID 37250266
- [Background] Grover N, Taneja R, Rashid Y, Shrivastava N. Nebulised fentanyl, dexmedetomidine and magnesium sulphate for attenuation of haemodynamic response to laryngoscopy and tracheal intubation: A double-blinded, randomised comparative study. Indian J Anaesth. 2023 Aug;67(8):730-735. doi: 10.4103/ija.ija_397_22. Epub 2023 Aug 15. PMID 37693019